CLINICAL TRIAL: NCT05825521
Title: Impact of Cerebral Ventricular Dilatations and Cerebrospinal Fluid Pulsations on Periventricular White Matter in Hydrocephalic Patients
Acronym: HYDRODIFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2021_843_0117
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hydrocephalus; Cerebral Ventricle; Cerebrospinal Fluid; White Matter Fiber
Keywords: Hydrocephalus; cerebral ventricles; cerebrospinal fluid; white matter fibers; functional biomarkers
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with hydrocephalus (Experimental): Age > 55, Ventricular dilation: Evans Index > 0.3; Patients with cognitive impairment, and gait disturbances and/or urinary incontinence or a combination of these three symptoms; Absence of other neurological diseases that could cause ventriculomegaly, information and non-opposition.
  Interventions: Other: MRI
- Controls (Active Comparator): Age ≥ 55; No ventricular dilation: Evans Index < 0.3; Individuals who have no neurological or psychiatric disease; No neurological deficit. No history of neurosurgery or head trauma; signed informed consent; affiliation to a social security scheme.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — During management, patients with hydrocephalus will be subjected to flow MRI and diffusion MRI. Flow parameters and diffusion parameters will be measured and compared to those found in control subjects receiving the same type of imaging

SUMMARY:
Hydrocephalus is characterized by excessive accumulation of cerebrospinal fluid (CSF) in the ventricles of the brain. One of the forms of hydrocephalus is called "normal pressure", although one of the main signs is precisely an alteration of the intracranial pressure (ICP), it is here called active hydrocephalus (HA). Although MRI is the reference radiological modality for the characterization of HA. The Evan's and DESH index are radiological diagnostic criteria based on the dilation and morphology of the CSF compartments. These morphological indices remain insensitive and specific. In recent years, advances in Phase Contrast (MRI-PC) and Diffusion (MRI-DTI) MRI have generated new biomarkers of brain viability. The aim of this study is to characterize by MRI the impact of hydrocephalus on brain fluids and tissues.

ELIGIBILITY:
Inclusion Criteria:

* For Patients with hydrocephalus:
* Age > 55,
* Ventricular dilation: Evans Index > 0.3;
* Patients with cognitive impairment, and gait disturbances and/or urinary incontinence or a combination of these three symptoms;
* Absence of other neurological diseases that could cause ventriculomegaly, information and non-opposition.
* For Controls:
* Age ≥ 55;
* No ventricular dilation: Evans Index < 0.3;
* Individuals who have no neurological or psychiatric disease;
* No neurological deficit.
* No history of neurosurgery or head trauma;
* signed informed consent;
* affiliation to a social security scheme.

Exclusion Criteria:

* All patients who have a neurological disease other than active hydrocephalus will be excluded;
* Individuals unable to sign or understand consent;
* Individuals with psychiatric, neurological or medical development;
* Individuals under treatment with psychoactive drugs;
* Individuals who cannot tolerate an MRI examination;
* Any individual with implant, pacemaker, prosthesis and ferromagnetic object

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Variation of MRI flow between both groups | 3 years
Variation of MRI diffusion between both groups | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No